CLINICAL TRIAL: NCT02328404
Title: The Effect of Vitamin D Supplementation on Chromium Serum Levels and Insulin Resistance Among Overweight Jordanian Women With Polycystic Ovary Syndrome in Irbid
Brief Title: The Effect of Vitamin D Supplementation Among Overweight Jordanian Women With Polycystic Ovary Syndrome (PCOS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hayat Pharmaceutical Co. PLC (Industry)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VitD31.0; 2013-003353-22 (EudraCT Number)
Record Dates: First submitted 2014-12-14; First posted 2014-12-31 (Estimated); Results first posted 2015-04-17 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-06

CONDITIONS: Polycystic Ovary Syndrome; Hypovitaminosis D
Keywords: Vitamin D; deficiency; hypovitaminosis D; Biodal; 25 hydroxy Vitamin D; 25hydroxyvitamin D; 25(OH)D; PCOS; insulin resistance; BMI; chromium levels; vitamin D 3; cholecalciferol; 50,000 IU
MeSH Terms: conditions — Polycystic Ovary Syndrome; Vitamin D Deficiency; Insulin Resistance | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitamin D3 (Biodal 50,000 IU) (Active Comparator): 50,000 IU Vitamin D3 tablet given orally once weekly for 3 months
  Interventions: Drug: 50,000 IU vitamin D3
- placebo (Placebo Comparator): Placebo tablet given orally once weekly for 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 50,000 IU vitamin D3 — Film-coated tablet Biodal 50,000 IU containing cholecalciferol 50,000 IU
  Other Names: Biodal 50,000 IU; cholecalciferol 50,000 IU
  Arms: vitamin D3 (Biodal 50,000 IU)
Drug: Placebo — Placebo film-coated tablet of Biodal 50,000 IU
  Other Names: Biodal 50,000IU
  Arms: placebo

SUMMARY:
This is a prospective double-blind, randomized, parallel-group, placebo-controlled trial designed to examine the effect of supplementation with 50,000 IU vitamin D3 for 3 months on Polycystic Ovary Syndrome (PCOS) prognosis, serum 25-Hydroxy Vitamin D (25(OH)D) level, serum chromium level, insulin resistance, and Body Mass Index (BMI), in 60 overweight Jordanian female patients diagnosed with PCOS and with hypovitaminosis D.

DETAILED DESCRIPTION:
This study is designed to assess the safety and efficacy of 50,000 IU vitamin D supplementation once weekly for 3 months on improvement in PCOS prognosis and improvement in serum 25(OH)D levels in 60 overweight Jordanian females (defined as having a BMI 25-30kg/m2), diagnosed with PCOS (based on Rotterdam criteria), and with hypovitaminosis D (defined as a serum 25(OH)D level < 20 ng/mL), compared with placebo.

Evaluation of the safety and efficacy of the dosing regimen will be conducted over 6 study visits during which clinical and biochemical signs of PCOS as well as serum 25(OH)D level, serum chromium level, insulin resistance, and BMI will be evaluated.

The measurements will be collected as follows : day (-7) during screening , Day (0) base line measurements , Day (30) , Day(60), Day (90), day (104).

ELIGIBILITY:
Inclusion Criteria:

* Female gender.
* Aged between 18 and 49 years old.
* Ethnic group (Caucasian, Middle-eastern).
* Overweight (BMI 25-30 kg^m2).
* Diagnosed with Polycystic ovary syndrome according to Rotterdam criteria (Rotterdam SHRE-ASRM Sponsored Polycystic ovary syndrome consensus workshop group, 2004).
* Diagnosed with hypovitaminosis D (serum 25(OH)D level < 20 ng/mL).
* Inadequate dietary intake of vitamin D (<600 IU/day or <15μg/day).
* Physical examination being assessed and accepted by the attending physician.
* Systolic blood pressure within the normal range (90-140 mmHg).
* Diastolic blood pressure within the normal range (60-90 mmHg).
* Heart rate within the normal range (60-100 BPM).
* Oral body temperature within the normal range (35.9 - 37.6 Cᵒ).
* Normal complete blood count , Liver Function enzymes test , Aspartate Transaminase (AST) , Alanine Transaminase (ALT) and Kidney function tests , Blood Urea Nitrogen (BUN) and Serum Creatinine (SrCr).
* Participant is willing and able to give informed consent for participation in the study.
* Able and willing to comply with all study requirements.

Exclusion Criteria:

* Female participants who are pregnant, lactating or planning pregnancy during the course of the study.
* Ethnic group: non Caucasian.
* Females aged <18 or >49 years old.
* Underweight, normal body weight ,Body Mass Index (BMI) < 25 kg^m2
* Obese or morbidly obese (BMI > 30 kg/m2)
* Diagnosis with type 1 or type 2 diabetes mellitus, hypothyroidism, hyperthyroidism, liver disease, renal dysfunction, cardiovascular diseases, androgen-secreting tumor, Cushing syndrome, congenital adrenal hyperplasia, hyperprolactinemia, and/or virilism.
* Known history or presence of food allergies or intolerance (e.g dairy products or gluten-containing foods), or any known condition that could interfere with the absorption, distribution, metabolism, or excretion of drugs.
* History of drug or alcohol abuse, smoking of 10 cigarettes or more (or equivalent) per day.
* Participants who took medications known to affect metabolic parameters, such as metformin and corticosteroid drugs, vitamin D and calcium.
* Adequate dietary intake of vitamin D (600 IU/day or 15μg/day or more).
* Participation in another clinical or bioequivalence study within 90 days prior to the start of this study period.
* Participants with abnormal Electrocardiogram (ECG).
* Participants with any abnormal laboratory results excluding [ 25(OH)D, Creatinine (Cr), Calcium (Ca), phosphorus (PO4), C-reactive protein(CRP) , triglyceride , High Density Lipoprotien Cholesterol (HDL-C), Low Density Lipoprotien Cholesterol (LDL-C), total cholesterol (TC)/HDL-C ratio, fasting insulin , fasting blood glucose, oral glucose tolerance test, impaired glucose tolerance, Progesterone, total testosterone, sex hormone binding globulin, parathyroid hormone and free androgen index].

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALA M ABU RUQAA, MSC PHARM, Study Director — HAYAT PHARMACEUTICAL INDUSTRIES CO. PLC
Locations (1):
- King Abdullah University Hospital, Irbid, Irbid Governorate, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Bayyari N, Al-Domi H, Zayed F, Hailat R, Eaton A. Androgens and hirsutism score of overweight women with polycystic ovary syndrome improved after vitamin D treatment: A randomized placebo controlled clinical trial. Clin Nutr. 2021 Mar;40(3):870-878. doi: 10.1016/j.clnu.2020.09.024. Epub 2020 Sep 24. PMID 33010974

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Random sample of women attending outpatient obstetrics and gynecology clinics in King Abdullah Hospital / Jordan University of Science and Technology
Pre-assignment Details: Approximately 120 women will be assessed for eligibility clinically, anthropometrically, dietary and biochemically.
  Women diagnosed with PCOS and vitamin D deficiency will be randomly divided into 2 groups
Groups:
- Vitamin D3 (Biodal 50,000IU): 50,000 IU vitamin D3 (Biodal 50,000IU) coated tablets by oral route
  50,000IU Vitamin D3: 50,000IU Vitamin D3 (Biodal 50,000IU ) once weekly for 3 months
- Placebo: placebo coated tablet by oral route
  placebo: placebo coated tablet by oral route
Period: Overall Study
Arm/Group | Vitamin D3 (Biodal 50,000IU) | Placebo
Started | 30 | 30
Completed | 29 | 29
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: Number of participants in each arm had been randomly allocated.
Groups:
- Placebo (Biodal 50,000IU Placebo): Placebo (Biodal 50,000IU Placebo tablets) coated tablets by oral route
  Placebo: 50,000IU Vitamin D3 placebo (Biodal 50,000IU placebo) once weekly for 3 months
- Total: Total of all reporting groups
Arm/Group | Vitamin D3 (Biodal 50,000IU) | Placebo (Biodal 50,000IU Placebo) | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Mean (Full Range); unit: years]
  Age | 23.56 [18 to 49] | 23.56 [18 to 49] | 23.56 [18 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 58
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Jordan | 29 | 29 | 58
Ultrasound Examination [Number; unit: participants]
  Both Overies are Normal | 0 | 0 | 0
  Left or Right is Normal | 0 | 0 | 0
  Both are Polycystic | 29 | 29 | 58
Hirsutism Score [Mean (Standard Deviation); unit: units on a scale] — The scale ranges between 0 and 36, where A score of 8 or higher was considered as androgen excess (Ferriman and Gallwey, 1961).
  Hirsutism score was assessed using self-administrated Ferriman-Gallwey scoring system (Ferriman and Gallwey, 1961). Each participant answered the hirsutism test with the help of a trained nurse who was working in the same clinic. The score of each body site may range between 0 (no excessive terminal hair growth) to 4 (extensive terminal hair growth).
  units on a scale | 16.5 (0.86) | 16.8 (1.19) | 16.65 (1.025)
25(OH)D Serum Level [Mean (Standard Deviation); unit: ng/ml] | 12.46 (3.29) | 12.37 (2.91) | 12.415 (3.08)
Progesterone Serum Level [Mean (Standard Deviation); unit: nmol/L] | 5.2 (1.86) | 10.7 (3.48) | 7.7 (2.67)
Total Testosteron Serum Level [Mean (Standard Deviation); unit: nmol/L] | 2.1 (0.17) | 1.8 (0.15) | 1.95 (0.16)
Chromium Serum Level [Mean (Standard Deviation); unit: ppm] | 0.29 (0.01) | 0.30 (0.01) | 0.295 (0.01)
Calcium Serum Level [Mean (Standard Deviation); unit: mmol/L] | 2.3 (0.02) | 2.3 (0.02) | 2.3 (0.02)
Phosphorus Serum Level [Mean (Standard Deviation); unit: nmol/L] | 1.1 (0.03) | 1.1 (0.02) | 1.1 (0.03)
Parathyroide Hormon Serum Level [Mean (Standard Deviation); unit: Pg/ml] | 65.3 (5.91) | 61.8 (4.54) | 63.55 (5.225)
Lipid Profile [Mean (Standard Deviation); unit: mmol/L]
  LDLC | 3.3 (0.15) | 3.4 (0.19) | 3.35 (0.17)
  HDL | 1.3 (0.06) | 1.3 (0.04) | 1.3 (0.05)
  Total Cholestrol | 5.3 (0.20) | 5.3 (0.26) | 5.3 (0.23)
TC / HDL-C Ratio [Mean (Standard Deviation); unit: Ratio] — This indicate the Total Cholesterol to High Density Lipoprotien ratio. An optimal ratio is between 3.5-to-1. A higher ratio means a higher risk of heart disease.
  Ratio | 4.3 (0.20) | 4.5 (0.26) | 4.4 (0.23)
Fasting Insulin Serum Level [Mean (Standard Deviation); unit: uU/ml] | 10.2 (1.23) | 9.8 (2.17) | 10.0 (3.4)
Fasting Blood Sugar Serum Level [Mean (Standard Deviation); unit: mmol/L] | 4.7 (0.07) | 4.9 (0.07) | 4.83 (0.04)
C-Reactive Protien Serum Level [Mean (Standard Deviation); unit: mg/L] | 6.6 (1.13) | 3.7 (0.69) | 5.15 (0.91)
Oral Glucose Tolerance Test (1st Hour) [Mean (Standard Deviation); unit: mmol/L] | 7.4 (0.33) | 7.7 (0.48) | 7.55 (0.41)
Sex Hormon Binding Globulin [Mean (Standard Deviation); unit: nmol/L] | 57.9 (9.29) | 111.2 (16.7) | 84.55 (13.00)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.33 (0.16) | 27.33 (0.30) | 27.33 (0.23)
Menstrual Cycle Regularity [Number; unit: participants]
  Regular | 3 | 4 | 7
  Irrigular | 26 | 25 | 51

OUTCOME MEASURES:

1. Primary Outcome: Ultrasound Examination of Number of Follicles and Ovarian Volume
Description: Evaluation of the efficacy of the dosing regimen as per the approved Summery of Product Characteristics (SmPC) (50,000 IU vitamin D3 once weekly for 3 months) on improvement in PCOS prognosis clinically using ultrasound examination.
  In this measure the reported results were the finding of the ultrasound examination after the course of the treatment /intervention as per the study protocol and reporting the numbers of patients with normal ovaries, One normal ovary and the other is polycystic or both ovaries are poly-cystic.
  An improvement in PCOS prognosis clinically by ultrasound examination is defined by:
  * decreasing the number of follicles to < 12 follicles measuring 2-9 mm in diameter
  * decreasing ovarian volume to < 10 cm3
Time Frame: 3 months
Population: The participants in the treatment and placebo groups will be classified into two categories of prognosis (improved and not improved) and will be analyzed using Chi-square test, if Chi-square is higher than 3.84 (df=1) it will be statistically significant (p-value</= 0.05)
Measure: Number; unit: participants
Arm/Group | Vitamin D3 (Biodal 50,000IU) | Placebo
Number analyzed (Participants) | 29 | 29
participants
  Both Normal | 7 | 0
  Left or Right Normal | 5 | 11
  Both Polycystic | 17 | 18
Statistical Analysis 1: Comparison: Vitamin D3 (Biodal 50,000IU) vs Placebo; The participants in the treatment and placebo groups will be classified into two categories of prognosis (improved and not improved) and will be analyzed using Chi-square test, if Chi-square is higher than 3.84 (df=1) it will be statistically significant (p-value</= 0.05); Test type: Superiority or Other; p = 0.001, Chi-squared; Fisher Exact test was used

2. Secondary Outcome: Serum 25-Hydroxy Vitamin D3 Level
Description: Evaluation of the Efficacy of the dose (50,000IU) and the dose regimen as per the approved SmPC on increase the level of serum 25(OH)D > 20 ng/ml by measuring of the serum 25(OH)D levels on 104 of the study period after 3 months treatment .
  In this measure , Serum 25-Hydroxy Vitamin D3 leveln in each arm were reported after completing the course of the treatment / intervention as per the study protocol. After which, the means were compared for statistical significance between the two groups / arms.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Vitamin D3 (Biodal 50,000IU) | Placebo
Number analyzed (Participants) | 29 | 29
ng/ml | 48.2 (2.03) | 11.8 (0.76)
Statistical Analysis 1: Comparison: Vitamin D3 (Biodal 50,000IU) vs Placebo; Both arms where evaluated at which paired t-test for the mean difference in the two arm was calculated . where the serum 25-OH Vit D3 was measured at 0 day time and after the end of the study. after that a paired t-test where applied for the difference for the 25-OH VitD3 levels between the two time points; Test type: Superiority or Other; p < 0.000, t-test, 2 sided — A P-value < 0.05 would be considered statistically significant

3. Secondary Outcome: Serum Chromium Concentration
Description: Evaluation of the Efficacy of the dose (50,000IU) and the dose regimen as per the approved SmPC on improving serum chromium level to be > 0.05 and < 0.5 ppm. which will be assessed by measuring serum chromium level before and after supplementation of Vitamin D3.
  In this measure , Serum chromium Concentration in each arm were reported after completing the course of the treatment / intervention as per the study protocol. After which, the means were compared for statistical significance between the two groups / arms.
  One of the clinical signs of improving PCOS prognosis is the improvement in serum chromium level . the results will be statistically analyzed using paired student t-test at 95% confidence interval (CI) for the difference of the means within and between the two groups will be calculated.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: ppm
Arm/Group | Vitamin D3 (Biodal 50,000IU) | Placebo
Number analyzed (Participants) | 29 | 29
ppm | 0.27 (0.01) | 0.27 (0.01)
Statistical Analysis 1: Comparison: Vitamin D3 (Biodal 50,000IU) vs Placebo; Test type: Superiority or Other; p = 0.67, t-test, 2 sided

4. Secondary Outcome: Serum Glucose Concentration in Oral Glucose Tolerance Test 1st hr After Treatment
Description: Evaluation of the Efficacy of the dose (50,000IU) and the dose regimen as per the approved SmPC on reduction of insulin resistance and improving insulin sensitivity measuring Oral Glucose Tolerance Test 1st hr after the treatment and to compare with same at baseline point within the time frame.
  In this measure , Serum Glucose Concentration in Oral Glucose Tolerance test in each arm were reported after completing the course of the treatment / intervention as per the study protocol (Treatment with either Biodal or Placebo for 3 months). After which, the means were compared for statistical significance between the two groups / arms.
  One of the clinical signs of improving PCOS prognosis is the improvement in insulin resistance by evaluating the results of Oral Glucose Tolerance Test 1st hr . the results will be statistically analyzed using paired student t-test at 95% confidence interval (CI).
Time Frame: 3 months
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Vitamin D3 (Biodal 50,000IU) | Placebo
Number analyzed (Participants) | 29 | 29
mmol/L | 6.9 (0.50) | 6.4 (0.54)
Statistical Analysis 1: Comparison: Vitamin D3 (Biodal 50,000IU) vs Placebo; Test type: Superiority or Other; p = 0.51, t-test, 2 sided

5. Secondary Outcome: Body Mass Index
Description: Evaluation of the Efficacy of the dose (50,000IU) and the dose regimen as per the approved SmPC on reduction of body mass index to be <25-30 kg/m^2.
  Evaluation of the Effectiveness of the dose (50,000IU) and the dose regimen as per the approved SmPC on reduction in Body Mass Index before and after the treatment. After which, the means were compared for statistical significance between the two groups / arms.
  In this measure , Body Mass Index in each arm were reported after completing the course of the treatment / intervention as per the study protocol (Treatment with either Biodal or Placebo for 3 months).
Time Frame: 3 months
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | Vitamin D3 (Biodal 50,000IU) | Placebo
Number analyzed (Participants) | 29 | 29
kg/m^2 | 25.6 (0.37) | 26.5 (0.37)
Statistical Analysis 1: Comparison: Vitamin D3 (Biodal 50,000IU) vs Placebo; Test type: Superiority or Other; p = 0.08, t-test, 2 sided

6. Secondary Outcome: Serum Parathyroid Hormone Concentration
Description: Evaluation of the Safety of the Dose and the Dose Regimen as Per the SmPC by measuring the change in the level of serum Serum Parathyroid Hormone (PTH) Concentration before and after the treatment and/or reporting any adverse events through the trial period.
  In this measure , Serum Parathyroid Hormone Concentration in each arm were reported after completing the course of the treatment / intervention as per the study protocol (Treatment with either Biodal or Placebo for 3 months). After which, the means were compared for statistical significance between the two groups / arms.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: Pg/ml
Groups:
- Vitamin D3 (Biodal 50,000IU): 50,000 IU vitamin D3 (Biodal 50,000IU) coated tablets by oral route
  50,000IU Vitamin D3: 50.000IU Vitamin D3 (Biodal 50,000IU ) once weekly for 3 months
Arm/Group | Vitamin D3 (Biodal 50,000IU) | Placebo
Number analyzed (Participants) | 29 | 29
Pg/ml | 39.1 (2.60) | 52.6 (4.18)
Statistical Analysis 1: Comparison: Vitamin D3 (Biodal 50,000IU) vs Placebo; Test type: Superiority or Other; p = 0.01, t-test, 2 sided

7. Primary Outcome: Menstrual Regularity
Description: Evaluation of the efficacy of the dosing regimen as per the approved SmPC (50,000 IU vitamin D3 once weekly for 3 months) on improvement in PCOS prognosis by assessment of menstrual regularity An improvement in PCOS prognosis by assessment of menstrual regularity is measured through improving progesterone level > 4 ng/mL.
  One of the clinical signs of improving PCOS prognosis is menstrual cycle regularity.
  In this measure ,the reported results consist of the number of volunteers/patients in each arm either with regular menstrual cycle or irregular menstrual cycle after completing the course of the treatment/ intervention as per the study protocol.
  The results will be statistically analyzed using paired student t-test and 95% confidence interval (CI) for the difference of the means within and between the two groups will be calculated.
Time Frame: 3 months
Measure: Number; unit: participants
Groups:
- Vitamin D3 (Biodal 50,000IU): 50,000 IU vitamin D3 (Biodal 50,000IU) coated tablets by oral route
  50.000IU Vitamin D3: 50,000IU Vitamin D3 (Biodal 50,000IU ) once weekly for 3 months
Arm/Group | Vitamin D3 (Biodal 50,000IU) | Placebo
Number analyzed (Participants) | 29 | 29
participants
  Regular | 27 | 4
  Irregular | 2 | 25
Statistical Analysis 1: Comparison: Vitamin D3 (Biodal 50,000IU) vs Placebo; Test type: Superiority or Other; p = 0.001, Chi-squared

8. Secondary Outcome: Serum Calcium Concentration
Description: Evaluation of the safety of the dose and the dose regimen as per the SmPC by measuring the change in the level of serum Calcium before and after the treatment and/or reporting it as adverse. event through the trial period. as the increase of Serum calcium concentration above the normal level is considered as adverse event for the intervention dose regimen of this study for the purpose of evaluating the safety.
  In this measure , Serum Calcium Concentration in each arm were reported after completing the course of the treatment / intervention as per the study protocol (Treatment with either Biodal or Placebo for 3 months). After which, the means were compared for statistical significance between the two groups / arms.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Vitamin D3 (Biodal 50,000IU) | Placebo
Number analyzed (Participants) | 29 | 29
mmol/L | 2.3 (0.02) | 2.3 (0.2)
Statistical Analysis 1: Comparison: Vitamin D3 (Biodal 50,000IU) vs Placebo; Test type: Superiority or Other; p = 0.89, t-test, 2 sided

9. Secondary Outcome: Serum Phosphorous Concentration
Description: Evaluation of the safety of the dose and the dose regimen as per the SmPC by measuring the change in the level of serum PO4 Concentration before and after the treatment and/or reporting as adverse event through the trial period.as the increase of Serum phosphoruse concentration above the normal level is considered as adverse event for the intervention dose regimen of this study for the purpose of evaluating the safety.
  In this measure , Serum Phosphorous Concentration in each arm were reported after completing the course of the treatment / intervention as per the study protocol (Treatment with either Biodal or Placebo for 3 months). After which, the means were compared for statistical significance between the two groups / arms.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Vitamin D3 (Biodal 50,000IU) | Placebo
Number analyzed (Participants) | 29 | 29
mmol/L | 1.2 (0.3) | 1.2 (0.2)
Statistical Analysis 1: Comparison: Vitamin D3 (Biodal 50,000IU) vs Placebo; Test type: Superiority or Other; p = 0.60, t-test, 2 sided

10. Primary Outcome: Hirsutism Score
Description: The scale ranges between 0 and 36, where A score of 8 or higher was considered as androgen excess (Ferriman and Gallwey, 1961).Evaluation of the Efficacy of the dose (50,000IU) and the dose regimen as per the approved SmPC on PCOS prognosis by evaluating Hirsutism Score.Hirsutism score was assessed using self-administrated Ferriman-Gallwey scoring system (Ferriman and Gallwey, 1961). Each participant answered the hirsutism test with the help of a trained nurse who was working in the same clinic. The score of each body site may range between 0 (no excessive terminal hair growth) to 4 (extensive terminal hair growth).
  In this measure , the hirsutism score were reported in each are after completing the course of treatment/ intervention as per the study protocol. after which, the means were compared for statistical significance between the two groups / arms.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: placebo coated tablet by oral route
  placebo (Biodal 50,000 IU): 50.000IU Vitamin D3 (Biodal 50.000IU ) placebo once weekly for 3 months
Arm/Group | Vitamin D3 (Biodal 50,000IU) | Placebo
Number analyzed (Participants) | 29 | 29
units on a scale | 11.5 (0.93) | 16.7 (1.21)
Statistical Analysis 1: Comparison: Vitamin D3 (Biodal 50,000IU) vs Placebo; Test type: Superiority or Other; p = 0.01, t-test, 2 sided

11. Secondary Outcome: Serum C-Reactive Protien Concentration
Description: Evaluation of the Efficacy of the Dose (50,000IU) and the Dose Regimen on inflammation by measuring reduction of the serum concentration of C-Reactive Protein before and after the treatment.
  In this measure , Serum C-Reactive Protien Concentration in each arm were reported after completing the course of the treatment / intervention as per the study protocol (Treatment with either Biodal or Placebo for 3 months). After which, the means were compared for statistical significance between the two groups / arms.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Vitamin D3 (Biodal 50,000IU) | Placebo
Number analyzed (Participants) | 29 | 29
mg/L | 5.4 (1.06) | 3.9 (1.17)
Statistical Analysis 1: Comparison: Vitamin D3 (Biodal 50,000IU) vs Placebo; Test type: Superiority or Other; p = 0.35, t-test, 2 sided

12. Primary Outcome: Serum Progesterone Level
Description: The results below show the Serum Progesterone level after treatment in each arm after completing the course of the treatment / intervention as per the study protocol.after which, the means were compared for statistical significance between the two groups / arms. After which, the means were compared for statistical significance between the two groups / arms.
  The evaluation of the Efficacy of the dose (50,000IU) and the dose regimen as per the approved SmPC on PCOS Prognosis by measuring Change in Serum Progesterone level.
  One of the clinical signs of improving PCOS prognosis is the change in progesterone level. the results will be statistically analyzed using paired student t-test at 95% confidence interval (CI) for the difference of the means within and between the two groups will be calculated.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Vitamin D3 (Biodal 50,000IU) | Placebo
Number analyzed (Participants) | 29 | 29
nmol/L | 5.8 (1.86) | 7.3 (2.42)
Statistical Analysis 1: Comparison: Vitamin D3 (Biodal 50,000IU) vs Placebo; Test type: Superiority or Other; p = 0.65, t-test, 2 sided

13. Primary Outcome: Total Testosterone Level
Description: Evaluation of the Efficacy of the dose (50,000IU) and the dose regimen as per the approved SmPC on PCOS Prognosis by measuring Change in Total Testosterone level before and after the treatment.
  In this measure , the Total Testosterone levels in each arm were reported after completing the course of the treatment / intervention as per the study protocol.
  One of the clinical signs of improving PCOS prognosis is the change in testosterone level. After which, the means were compared for statistical significance between the two groups / arms.
  the results will be statistically analyzed using paired student t-test at 95% confidence interval (CI) for the difference of the means within and between the two groups will be calculated.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Vitamin D3 (Biodal 50,000IU) | Placebo
Number analyzed (Participants) | 29 | 29
nmol/L | 1.6 (0.17) | 1.9 (0.1)
Statistical Analysis 1: Comparison: Vitamin D3 (Biodal 50,000IU) vs Placebo; Test type: Superiority or Other; p = 0.25, t-test, 2 sided

14. Primary Outcome: Free Androgen Index
Description: Free Androgen Index is calculated as the ratio of total testosterone to sex hormone binding globulin (SHBG).
  In this measure , the Free Androgen Index in each arm were reported after completing the course of the treatment / intervention as per the study protocol. After which, the means were compared for statistical significance between the two groups / arms.
  Improvement assessment of PCOS Prognosis by evaluating the change in Free Androgen Index.
  One of the clinical signs of improving PCOS prognosis is the change in FAI. the results will be statistically analyzed using Wilcoxon (Mann- Whitney) method at 95% confidence interval (CI) for the difference of the means within and between the two groups will be calculated.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Vitamin D3 (Biodal 50,000IU) | Placebo
Number analyzed (Participants) | 29 | 29
Ratio | 4.5 (0.93) | 4.4 (1.10)
Statistical Analysis 1: Comparison: Vitamin D3 (Biodal 50,000IU) vs Placebo; Test type: Superiority or Other; p = 0.04, Wilcoxon (Mann-Whitney)

15. Primary Outcome: Sex Hormone Binding Globulin Concentration
Description: Evaluation of Biodal 50,000 IU on improvement of PCOS Prognosis by comparing the Sex Hormone Binding Globulin concentrations in both groups/arms.
  One of the clinical signs of improving PCOS prognosis is the change in the Sex Hormone Binding Globulin Concentration.
  In this measure , the Sex Hormone Binding Globulin Concentration in each arm were reported after completing the course of the treatment / intervention as per the study protocol. After which, the means were compared for statistical significance between the two groups / arms.
  The results will be statistically analyzed using Wilcoxon (Mann-Whiteny) method at 95% confidence interval (CI) for the difference of the means within and between the two groups will be calculated.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Vitamin D3 (Biodal 50,000IU) | Placebo
Number analyzed (Participants) | 29 | 29
nmol/L | 85.9 (15.19) | 100.6 (15.8)
Statistical Analysis 1: Comparison: Vitamin D3 (Biodal 50,000IU) vs Placebo; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Baseline, 3 months
Description: Vitamin D supplementation for vitamin D deficient (<20 ng/ml) women with 50,000 IU/week for 12 weeks did not lead to any side effects.
Arm/Group | Vitamin D3 (Biodal 50,000IU) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 1/30 | 1/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D3 (Biodal 50,000IU) (N=30) | Placebo (N=30)
In-compliance , Withdral (Social circumstances) | 1 (1) | 1 (1) — One Volunteer was dropped out due to in-compliance / Not responding to phone call. One Volunteer had withdrawn due to long term travel outside the country after starting the study

LIMITATIONS AND CAVEATS:
* The study was conducted only in the north of Jordan
* Body composition was measured by bioelectrical impedance
* Insulin resistance was assessed using the indirect method of assessment (HOMA)
* The study was done exclusively on overweight women

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No